CLINICAL TRIAL: NCT00022659
Title: A Phase II Evaluation of Bevacizumab (Anti-VEGF Humanized Monoclonal Antibody) (NSC #704865) in the Treatment of Persistent or Recurrent Epithelial Ovarian or Primary Peritoneal Carcinoma
Brief Title: Bevacizumab in Treating Patients With Persistent or Recurrent Ovarian Epithelial Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02400; NCI-2012-02400 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000068839; GOG-0170D (Other: Gynecologic Oncology Group); GOG-0170D (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer; Stage IV Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Bevacizumab

ARMS (1):
- Treatment (bevacizumab) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is to see if bevacizumab works in treating patients who have persistent or recurrent ovarian epithelial cancer or primary peritoneal cancer. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the 6-month progression-free survival of patients with persistent or recurrent ovarian epithelial or primary peritoneal cancer treated with bevacizumab.

II. Determine the nature and degree of toxicity of this drug in these patients. III. Determine the progression-free and overall survival of patients treated with this drug.

IV. Determine the frequency of clinical response in patients treated with this drug.

V. Determine the effect of this drug on initial performance status, age, and mucinous or clear cell histology in these patients.

VI. Correlate biological and imaging markers with 6-month progression-free survival of patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian epithelial or primary peritoneal carcinoma

  * Recurrent or persistent after initial standard surgery or chemotherapy
  * Incurable with standard surgery, chemotherapy, or radiotherapy
* At least 1 unidimensionally measurable target lesion

  * At least 20 mm by conventional techniques
  * At least 10 mm by spiral CT scan
  * Outside the area of prior radiotherapy
* Accessible to guided core needle biopsy
* Received 1 prior platinum-based chemotherapy regimen (e.g., carboplatin, cisplatin, or another organoplatinum compound) for primary disease

  * May have included high-dose therapy, consolidation, or extended therapy administered after surgical or non-surgical assessment
  * Patients with only 1 prior platinum-based chemotherapy regimen must have an initial treatment-free interval of less than 12 months
  * Patients with an initial treatment-free interval of more than 12 months must have progressive disease after prior platinum-based chemotherapy regimen as second-line therapy
* No tumors involving major blood vessels
* No evidence of CNS disease (primary brain tumor or brain metastases) within the past 5 years
* Ineligible for higher priority Gynecologic Oncology Group (GOG) protocols (i.e., active phase III GOG protocols for the same patient population)
* Performance status - GOG 0-2 (patients who have received 1 prior regimen)
* Performance status - GOG 0-1 (patients who have received 2 prior regimens)
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No known bleeding disorder or coagulopathy
* No active bleeding
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* serum glutamate oxaloacetate transaminase (SGOT) ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* PT (INR) ≤ 1.5 (INR 2-3 if on stable dose of therapeutic warfarin or low molecular weight heparin)
* Partial thromboplastin time (PTT) < 1.2 times control
* Creatinine ≤ 1.5 times ULN
* Creatinine clearance > 60 mL/min
* No proteinuria, as indicated by 1 of the following:

  * Negative urine dipstick
  * Urine protein < 30 mg/dL
  * Urine protein < 1,000 mg on 24-hour urine collection
* No clinically significant cardiovascular disease, including any of the following:

  * Uncontrolled hypertension
  * Myocardial infarction within the past 6 months
  * Unstable angina within the past 6 months
  * New York Heart Association class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Peripheral vascular disease ≥ grade 2
* No stroke within the past 5 years
* No pathologic condition that carries a high risk of bleeding
* No significant traumatic injury within the past 28 days
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No uncontrolled seizures within the past 5 years
* No neuropathy (motor and sensory) ≥ grade 2
* No serious non-healing wound, ulcer, or bone fracture
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* No active infection requiring parenteral antibiotics
* No known claustrophobia that would preclude MRI tolerance
* No ferromagnetic implants or pacers
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study treatment
* At least 3 weeks since prior immunologic therapy directed at malignancy
* No prior bevacizumab
* No other concurrent immunotherapy directed at malignancy
* One additional prior cytotoxic regimen for recurrent or persistent disease allowed
* No prior non-cytotoxic chemotherapy for recurrent or persistent disease
* No concurrent chemotherapy directed at malignancy
* At least 1 week since prior hormonal therapy directed at malignancy
* No concurrent hormonal therapy directed at malignancy
* Concurrent hormone replacement therapy allowed
* Recovered from prior radiotherapy
* No concurrent radiotherapy directed at malignancy
* At least 28 days since prior major surgery or open biopsy and recovered
* At least 7 days since prior core biopsy or placement of vascular access device
* No anticipated need for major surgical procedure during study participation
* At least 3 weeks since other prior therapy directed at malignancy
* No prior anticancer therapy that would preclude study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2002-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Burger, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 4/29/2002 and closed to accrual on 8/25/2004 (suspended from 10/6/2003 to 12/1/2003).
Groups:
- Bevacizumab: Bevacizumab 15 mg/kg IV, every 3 weeks (one cycle) until disease progression or adverse effects prohibit further therapy
Period: Overall Study
Arm/Group | Bevacizumab
Started | 64
Completed | 62 (Eligible and treated patients.)
Not Completed | 2
Not completed — Ineligible: wrong primary | 1
Not completed — Never treated | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (12.5)
Age, Customized [Number; unit: participants]
  10-19 years | 1
  20-29 years | 1
  30-39 years | 3
  40-49 years | 13
  50-59 years | 21
  60-69 years | 13
  70-79 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 62
Histologic Type [Number; unit: participants]
  Adenocarcinoma, Unspecified | 1
  Clear Cell Carcinoma | 2
  Endometrioid Adenocarcinoma | 2
  Mixed Epithelial Carcinoma | 6
  Serous Adenocarcinoma | 51

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 6 Months
Description: Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions.
Time Frame: Every other cycle for 6 months.
Population: Eligible and treated patients.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 62
percentage of participants | 40.3 [29.8 to 53.6]

2. Primary Outcome: Tumor Response
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: Every other cycle for the first 6 months; then every 3 months x 2 ; then every 6 months thereafter for up to 5 years.
Population: Eligible and treated patients.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 62
percentage of participants | 21 [12.6 to 31.3]

3. Primary Outcome: Number of Participants and Degree of Toxicity of Bevacizumab in This Cohort of Patients as Assessed by CTC.
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment, up to 5 years.
Population: Eligible and evaluable patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 1 (CTCAE v 2.0): Number of patients who experienced a grade 1 event using Common Toxicity Criteria version 2.0
- Grade 2 (CTCAE v 2.0): Number of patients who experienced a grade 2 event using Common Toxicity Criteria version 2.0
- Grade 3 (CTCAE v 2.0): Number of patients who experienced a grade 3 event using Common Toxicity Criteria version 2.0
- Grade 4 (CTCAE v 2.0): Number of patients who experienced a grade 4 event using Common Toxicity Criteria version 2.0
Arm/Group | Grade 1 (CTCAE v 2.0) | Grade 2 (CTCAE v 2.0) | Grade 3 (CTCAE v 2.0) | Grade 4 (CTCAE v 2.0)
Number analyzed (Participants) | 62 | 62 | 62 | 62
Participants
  Leukopenia | 18 | 0 | 0 | 0
  Thrombocytopenia | 6 | 0 | 0 | 0
  Neutropenia | 6 | 3 | 0 | 0
  Anemia | 18 | 1 | 0 | 0
  Hematologic | 2 | 1 | 1 | 0
  Allergy | 3 | 0 | 2 | 0
  Hearing | 2 | 0 | 0 | 0
  Cardiovascular | 12 | 1 | 7 | 1
  Coagulation | 9 | 2 | 1 | 0
  Constitutional | 22 | 6 | 1 | 0
  Dermatologic | 10 | 2 | 0 | 0
  Endocrine | 3 | 0 | 0 | 0
  Gastrointestinal | 26 | 6 | 3 | 1
  Genitourinary/Renal | 5 | 14 | 0 | 1
  Hemorrhage | 14 | 0 | 0 | 0
  Hepatic | 19 | 2 | 1 | 0
  Infection | 3 | 6 | 0 | 0
  Lymphatics | 2 | 0 | 0 | 0
  Musculoskeletal | 4 | 1 | 0 | 0
  Metabolic | 17 | 0 | 0 | 0
  Neurologic | 16 | 1 | 0 | 0
  Ocular | 2 | 1 | 0 | 0
  Pain | 26 | 6 | 3 | 0
  Pulmonary | 6 | 6 | 1 | 0
  Sexual/Reproductive | 2 | 0 | 0 | 0

4. Secondary Outcome: Overall Survival
Description: The observed length of life from entry into the study to death or the date of last contact.
Time Frame: From study entry to death or last contact, up to 5 years.
Population: Eligible and treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 62
months | 16.9 [11.8 to 27.2]

5. Secondary Outcome: Duration of Progression-free Survival
Description: as for outcome 1
Time Frame: Every other cycle for the first 6 months; then every 3 months x 2 ; then every 6 months therafter for up to 5 years.
Population: Eligible and treated patients
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 62
months | 4.7 [2.7 to 12.9]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adverse Events (SAEs) up to 5 years after stopping study treatment
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 26/62
Other Adverse Events (participants affected / at risk) | 62/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=62)
Allergic Reaction (Immune system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Hematologic Other (Blood and lymphatic system disorders) | 1
Edema (Cardiac disorders) | 1
Thrombosis Embolism (Cardiac disorders) | 2
Ischemia/Cardiac Infarction (Cardiac disorders) | 1
Partial Thromboplastin Time (Vascular disorders) | 1
Weight Gain(No Vod) (General disorders) | 1
Flushing (Skin and subcutaneous tissue disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Vomitting (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Gi Other (Gastrointestinal disorders) | 2
Melena/Gi Bleeding (Vascular disorders) | 1
Abdominal Pain (General disorders) | 1
Pain Tumor (General disorders) | 1
Voice Changes/Stridor/Larynx (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=62)
Allergic Rhinitis (Immune system disorders) | 8
Allergic Reaction (Immune system disorders) | 3
Inner Ear/Hearing (Ear and labyrinth disorders) | 4
Middle Ear/Hearing (Ear and labyrinth disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Lymphopenia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 22
Transfusion Prbc's (Blood and lymphatic system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 30
Hematologic Other (Blood and lymphatic system disorders) | 1
Conduction Abnorm Atrioventricular Block (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 3
Sinus Tachycardia (Cardiac disorders) | 4
Arrhythmia Super Ventricular (Cardiac disorders) | 1
Phlebitis Superficial (Cardiac disorders) | 1
Sinus Bradycardia (Cardiac disorders) | 1
Edema (Cardiac disorders) | 10
Thrombosis Embolism (Cardiac disorders) | 3
Hypertension (Cardiac disorders) | 18
Palpitations (Cardiac disorders) | 1
Ischemia/Cardiac Infarction (Cardiac disorders) | 1
Prothrombin Time (Vascular disorders) | 1
Coagulation Other (Vascular disorders) | 8
Partial Thromboplastin Time (Vascular disorders) | 10
Fever(No Neutropenia) (General disorders) | 5
Weight Loss (General disorders) | 8
Rigors Chills (General disorders) | 3
Weight Gain(No Vod) (General disorders) | 2
Sweating (General disorders) | 3
Fatigue (General disorders) | 40
Pruritis (Skin and subcutaneous tissue disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 6
Rash Desquamation (Skin and subcutaneous tissue disorders) | 7
Skin Other (Skin and subcutaneous tissue disorders) | 1
Nail Changes (Skin and subcutaneous tissue disorders) | 3
Pigmentation Changes (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 1
Bruising (Skin and subcutaneous tissue disorders) | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Hypothyroidism (Endocrine disorders) | 2
Hot Flashes/Flushes (Endocrine disorders) | 8
Anorexia (Gastrointestinal disorders) | 12
Flatulence (Gastrointestinal disorders) | 4
Diarrhea With Colostomy (Gastrointestinal disorders) | 1
Mouth Dryness (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 3
Ascites Non-Malignant (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Dyspepsia/Heartburn (Gastrointestinal disorders) | 10
Taste Disturbance (Gastrointestinal disorders) | 1
Dysphagia Esophagitis Odynophagia (Gastrointestinal disorders) | 4
Diarrhea Without Colostomy (Gastrointestinal disorders) | 18
Constipation (Gastrointestinal disorders) | 24
Stomatitis/Pharyngitis (Gastrointestinal disorders) | 11
Dehydration (Gastrointestinal disorders) | 3
Vomitting (Gastrointestinal disorders) | 21
Nausea (Gastrointestinal disorders) | 27
Gi Other (Gastrointestinal disorders) | 13
Hemorrhage Other (Vascular disorders) | 4
Rectal Bleeding/Hematochezia (Vascular disorders) | 4
Epistaxis (Vascular disorders) | 6
Melena/Gi Bleeding (Vascular disorders) | 1
Hemorrhage Without Grade 3/4 Thrombocytopenia (Vascular disorders) | 2
Vaginal Bleeding (Vascular disorders) | 3
Hematuria No Vaginal Bleeding (Vascular disorders) | 4
Ggt(Gamma-Glutamyltranspeptidase) (Hepatobiliary disorders) | 1
Hepatic Other (Hepatobiliary disorders) | 2
Hypoalbuminemia (Hepatobiliary disorders) | 12
Sgot(Alt) (Hepatobiliary disorders) | 11
Sgot(Ast) (Hepatobiliary disorders) | 19
Alkaline Phosphatase (Hepatobiliary disorders) | 17
Bilirubin (Hepatobiliary disorders) | 4
Infection Without Neutropenia (Infections and infestations) | 26
Lymphatics Other (Blood and lymphatic system disorders) | 1
Lymphatics (Blood and lymphatic system disorders) | 2
Alkalosis (Metabolism and nutrition disorders) | 1
Hypercholesterolemia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 8
Metabolic Other (Metabolism and nutrition disorders) | 14
Hyponatremia (Metabolism and nutrition disorders) | 11
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypertyiglyceridemia (Metabolism and nutrition disorders) | 3
Bicarbonate (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 16
Hypoglycemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hypomagnesmia (Metabolism and nutrition disorders) | 12
Musculoskeletal Other (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 7
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4
Extrapyramidal (Nervous system disorders) | 1
Depressed Level Of Consciousness (Nervous system disorders) | 1
Vertigo (Nervous system disorders) | 1
Mood Alteration Anxeity/Agitation (Nervous system disorders) | 16
Memory Loss (Nervous system disorders) | 2
Insomnia (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 9
Mood Alteration Depression (Nervous system disorders) | 9
Neuropathy Sensor (Nervous system disorders) | 15
Pyramidal Tract Dysfunction (Nervous system disorders) | 1
Glaucoma (Eye disorders) | 1
Ocular Other (Eye disorders) | 2
Tearing (Eye disorders) | 1
Dry Eye (Eye disorders) | 2
Cataract (Eye disorders) | 3
Vision Blurres (Eye disorders) | 2
Abdominal Pain (General disorders) | 29
Pain Other (General disorders) | 14
Pain Tumor (General disorders) | 5
Pleuritic Pain (General disorders) | 2
Neuropathic Pain (General disorders) | 1
Earache (General disorders) | 1
Dyspareunia (General disorders) | 2
Headache (General disorders) | 19
Pelvic Pain (General disorders) | 7
Chest Pain (General disorders) | 6
Bone Pain (General disorders) | 3
Arthralgia (General disorders) | 14
Myalgia (General disorders) | 17
Pain Rectal/Perirectal (General disorders) | 1
Voice Changes/Stridor/Larynx (Respiratory, thoracic and mediastinal disorders) | 7
Pulmonary Other (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Ards (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16
Urinary Frequency/Urgency (Renal and urinary disorders) | 5
Dysuria (Renal and urinary disorders) | 5
Creatinine (Renal and urinary disorders) | 4
Renal/Gu Other (Renal and urinary disorders) | 3
Vaginitis No Infection (Renal and urinary disorders) | 4
Ureteral Obstruction (Renal and urinary disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Hemoglobinuria (Renal and urinary disorders) | 1
Bladder Spasms (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 22
Vaginal Dryness (Reproductive system and breast disorders) | 3
Libido (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less